CLINICAL TRIAL: NCT00006502
Title: Myocardial Perfusion, Risk Factors, and Coronary Calcium
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 943; R01HL065580 (NIH)
Record Dates: First submitted 2000-11-16; First posted 2000-11-17 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2005-07

CONDITIONS: Cardiovascular Diseases; Coronary Arteriosclerosis; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease; Heart Diseases

SUMMARY:
To determine whether an impairment of myocardial perfusion reserve is an early indicator of coronary artery disease.

DETAILED DESCRIPTION:
BACKGROUND:

Impairment of coronary vasofunction is believed to be one of the earliest manifestations of coronary heart disease (CHD). The impact of risk factors such as elevated cholesterol levels, diabetes, hypertension, and smoking on the coronary microcirculation remains largely unknown.

DESIGN NARRATIVE:

The cross-sectional study will determine whether an impairment of the myocardial perfusion reserve provides a marker of coronary heart disease (CHD) by comparing it to other novel measures of subclinical vascular disease, and by testing its association with risk factors for CHD. The study is ancillary to the Multi-Ethnic Study of Atherosclerosis ("MESA"), which is an NHLBI funded, prospective observational study of the characteristics of subclinical cardiovascular disease, i.e. disease detected non-invasively before it has produced signs and symptoms. In MESA new measures of subclinical disease such as coronary artery calcium and impaired brachial artery reactivity are to be examined to investigate their relationships to well-established risk factors and clinical events. Myocardial perfusion reserve (MPR)is a useful measure of coronary vasofunction that should be included in an evaluation of new measures of subclinical disease. An impaired MPR appears to be a specific early indicator of the functional impairment of the microcirculation in patients with risk factors for coronary artery disease. Magnetic resonance imaging (MRI) will be used as an advanced, quantitative imaging modality to determine in short (20 minute) exams the myocardial perfusion reserve in a group of 400 MESA participants. The study tests the hypothesis that impaired myocardial perfusion reserve indicates the presence of subclinical coronary atherosclerosis and coronary microvascular disease.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-09; Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jerosch-Herold — University of Minnesota

REFERENCES:
- [Background] Jerosch-Herold M, Swingen C, Seethamraju RT. Myocardial blood flow quantification with MRI by model-independent deconvolution. Med Phys. 2002 May;29(5):886-97. doi: 10.1118/1.1473135. PMID 12033585
- [Background] Swingen C, Seethamraju RT, Jerosch-Herold M. An approach to the three-dimensional display of left ventricular function and viability using MRI. Int J Cardiovasc Imaging. 2003 Aug;19(4):325-36. doi: 10.1023/a:1025450211508. PMID 14598902
- [Background] Jerosch-Herold M, Hu X, Murthy NS, Rickers C, Stillman AE. Magnetic resonance imaging of myocardial contrast enhancement with MS-325 and its relation to myocardial blood flow and the perfusion reserve. J Magn Reson Imaging. 2003 Nov;18(5):544-54. doi: 10.1002/jmri.10384. PMID 14579397
- [Background] Swingen CM, Seethamraju RT, Jerosch-Herold M. Feedback-assisted three-dimensional reconstruction of the left ventricle with MRI. J Magn Reson Imaging. 2003 May;17(5):528-37. doi: 10.1002/jmri.10290. PMID 12720262
- [Background] Jerosch-Herold M, Seethamraju RT, Swingen CM, Wilke NM, Stillman AE. Analysis of myocardial perfusion MRI. J Magn Reson Imaging. 2004 Jun;19(6):758-70. doi: 10.1002/jmri.20065. PMID 15170782